CLINICAL TRIAL: NCT05524454
Title: Evaluation of a Cone-beam CT Scanner for Image Guided Radiotherapy (CONFIGURE)
Brief Title: Evaluation of a Cone-beam CT Scanner for Image Guided Radiotherapy
Acronym: CONFIGURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VAR-2022-04
Record Dates: First submitted 2022-08-29; First posted 2022-09-01 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer; Lung Cancer; Breast Cancer; Abdominal Cancer; Pelvic Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Breast Neoplasms; Pelvic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-site study designed to generate data describing the quality and applicability of a novel on-couch CBCT imaging system for anatomy visualization and radiation treatment dosimetry planning.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Novel CBCT Imaging (Experimental): All subjects undergo one additional imaging session with the novel CBCT imaging system.
  Interventions: Device: Novel CBCT Imaging

INTERVENTIONS:
Device: Novel CBCT Imaging — One or two CBCT images are acquired on the novel CBCT imaging system.

SUMMARY:
This is a feasibility study investigating the image quality of a new, high-performance cone beam CT (CBCT) used for on-couch imaging during radiotherapy treatments.

DETAILED DESCRIPTION:
This study will examine the image quality generated by a new cone-beam CT (CBCT) imaging system integrated into an external beam radiation treatment delivery platform. Normally, CBCT images are acquired at the start of a daily radiation delivery treatment to align the patient with the images that were used to generate their radiation treatment plan. This alignment increases the precision of radiation delivery. This study will assess whether the improvements in image quality expected from the novel CBCT imaging system are sufficient for the images to be used for more than just patient alignment.

The study will enroll patients who will be treated with external beam radiation therapy for the following conditions: head and neck cancers, stage I lung cancer, stage II to IV lung cancer, cancer in the left breast, tumors in the abdomen, and tumors in the pelvic region. Each patient will undergo one additional imaging session with the novel CBCT imaging system during which 1 or 2 CBCT images will be acquired. The number of novel CBCT images acquired depends on the location and type of the patient's tumor. The additional imaging session will occur on the same day as one of the patient's scheduled treatment delivery sessions to minimize impact on the patient's schedule.

The patient's cancer treatment will not be affected by participation in this study. The methodology for the subject's treatment setup, CT simulation, treatment planning, image guidance and treatment delivery will be determined by the subject's treatment team.

The images acquired by the novel CBCT imaging system will be compared to standard CBCT images acquired as part of the patient's treatment and to the CT simulation images used to define the patient's radiation treatment plan.

ELIGIBILITY:
Inclusion Criteria:

* The patient will be treated with external beam photon radiotherapy at Maastro for head-and-neck cancer, stage I lung cancer, stage II-IV lung cancer, left breast cancer, or tumours in the abdominal or pelvic region.
* Age ≥ 18 years
* Ability to understand the requirements of the study and to give written informed consent, as determined by the treating physician
* Provision of written informed consent

Exclusion Criteria:

* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht Radiation Oncology, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Novel CBCT Imaging
Started | 41
Completed | 40
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are provided for study participants who had study imaging performed.
Arm/Group | Novel CBCT Imaging
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 67 [45 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] — Population: Height and/or weight values were not available for 2 study participants.
  kg/m^2
    number analyzed (Participants) | 38
    (all) | 26.4 [18.2 to 35.8]

OUTCOME MEASURES:

1. Primary Outcome: Image Quality
Description: For this objective, the image noise level was evaluated in regions of interest representing different tissue types (muscle and fat) in both CT simulation images and HyperSight CBCT images. Image noise is the variation in image intensity, which is measured in Hounsfield Units (HU), in a region that should have uniform intensity without the presence of noise. Image noise is measured as the standard deviation of HU within the defined regions of interest. Higher noise values indicate poorer image quality. HyperSight images can be reconstructed from raw data using different reconstruction algorithms. For this analysis, both the standard Feldkamp-Davis-Kress (FDK) algorithm and an iterative metal artifact reduction (MAR) algorithm were evaluated.
Time Frame: Within 1 month from the start of treatment
Population: Images were analyzed according to the anatomical region being imaged. As of the last date of publication to ClinicalTrials.gov, only data for the 7 Head/Neck participants were available.
Measure: Median (Full Range); unit: standard deviation of HU values
Groups:
- Head/Neck Imaging: Evaluation of images of study participants treated for head/neck cancer.
Arm/Group | Head/Neck Imaging
Number analyzed (Participants) | 7
standard deviation of HU values
  Noise in muscle for planning CT | 6.6 [4.2 to 8.3]
  Noise in muscle for HyperSight MAR | 9.8 [3.9 to 14.9]
  Noise in muscle for HyperSight FDK | 11.2 [8.8 to 27.4]
  Noise in fat for planning CT | 8.9 [4.6 to 13.1]
  Noise in fat for HyperSight MAR | 7.1 [3.6 to 15.3]
  Noise in fat for HyperSight FDK | 7.6 [3.1 to 23.0]

2. Secondary Outcome: Accuracy of Radiation Dose Calculation on HyperSight CBCT
Description: The accuracy of dose calculation on HyperSight CBCT was evaluated by re-calculating a participant's clinical treatment plan on one of their HyperSight images and comparing the doses delivered to target structures and organs at risk (OARs). The lower the difference in dose metrics between a HyperSight CBCT-based plan and a CT simulation-based plan, the more accurate the dose calculation on HyperSight CBCT.
  Both the maximum dose delivered to OARs and the mean dose delivered to OARs were compared between HyperSight-based plans and CT simulation-based plans. We report the worst overall accuracy, i.e. maximum difference in dose metrics across all OARs from across all patients. Similarly, the maximum dose delivered to the target, the mean dose delivered to the target and the minimum dose delivered to 95% of the target were compared between HyperSight CBCT-based plans and CT simulation-based plans. We report here the maximum difference across all dose metrics from across all patients.
Time Frame: Within 1 month from the start of treatment
Population: Dose calculation accuracy was analyzed according to the anatomical region being imaged. As of the last date of publication to ClinicalTrials.gov, only data for the 7 Head/Neck participants were available.
Measure: Number; unit: Gy
Arm/Group | Head/Neck Imaging
Number analyzed (Participants) | 7
Gy
  Max difference in OAR DVH metrics between HyperSight MAR and CT simulation across all subjects. | 1.1
  Max difference in target DVH metrics between HyperSight MAR and CT simulation across all subjects. | 6.5

3. Secondary Outcome: Qualitative Assessment of Novel CBCT Images for Contouring Organs at Risk
Description: CT simulation images and HyperSight CBCTs from subjects were randomly presented to expert reviewers, who were blinded to the type of image they were looking at and who were asked to rate their confidence level for contouring organs at risk (OARs) on the images using a 5-point Likert scale (very high, high, moderate, low, very low). The percentage of times that a reviewer rated their confidence level for contouring OARs on HyperSight CBCT as moderate, high, or very high was recorded. A higher percentage means a more favorable assessment for OAR contouring on HyperSight CBCT. The percentage of times the reviewer's confidence level for contouring on a HyperSight CBCT was equal to or higher than their confidence level on the corresponding CT simulation image was also recorded, where again a higher percentage means a better assessment for OAR contouring on HyperSight CBCT. The HyperSight iterative metal artifact reconstruction (MAR) algorithm was used in this analysis.
Time Frame: Within 1 month from the start of treatment
Population: Images were assessed according to the anatomical region being imaged. As of the last date of publication to ClinicalTrials.gov, only data for the 7 Head/Neck participants were available. Seven observers evaluated two image series - CT simulation images and HyperSight CBCT - from each study participant.
Measure: Number; unit: % evaluations
Units Other Than Participants: Evaluations
Groups:
- Head/Neck Images: Evaluation of images of study participants treated for head/neck cancer.
Arm/Group | Head/Neck Images
Number analyzed (Participants) | 7
Number analyzed (Evaluations) | 98
% evaluations
  % evaluations OAR contouring confidence on HyperSight MAR was equal or higher than on CT simulation | 47
  Percentage of moderate, high, or very high confidence in contouring OARs on HyperSight | 70

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time a subject consented to participate in the study to the end of their radiation therapy treatment, or to the end of their participation in the study, whichever came first. The adverse event assessment period typically was from 2-6 weeks, depending on the duration of the participant's radiation treatment.
Description: Only adverse events that were Possibly, Probably, or Definitely attributable to HyperSight imaging were reported.
Arm/Group | Novel CBCT Imaging
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT05524454/Prot_SAP_000.pdf